CLINICAL TRIAL: NCT05823337
Title: Evaluation of the Relationship Between Serum Selenium Level and Glycemic Control in Pregnant Patients*
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ece Yigit, Ass.prof. Ece YİĞİT, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: gdmselenyum*
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Gestational Diabetes; Pregnancy Related
Keywords: selenium; gestational diabetes mellitus; glycemic control
MeSH Terms: conditions — Diabetes, Gestational | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- only given diet therapy (Active Comparator): only diet theraphy
  Interventions: Dietary Supplement: only diet
- given diet therapy and selenium (Experimental): diet theraphy and 200 mcg selenium
  Interventions: Dietary Supplement: selenium+ diet

INTERVENTIONS:
Dietary Supplement: selenium+ diet — Selenium functions as an active site component of an antioxidant enzyme, glutathione peroxidase, and helps scavenge free radicals.
  Other Names: diet
  Arms: given diet therapy and selenium
Dietary Supplement: only diet — diet suitable for pregnancy
  Arms: only given diet therapy

SUMMARY:
Gestational diabetes mellitus (GDM) occurs in approximately 15% of all pregnancies worldwide.GDM can lead to the development of type 2 diabetes mellitus (T2DM) later in a woman's life. Babies of mothers with GDM have a greater risk of developing T2DM and cardiovascular disease than infants of women without GDM. The degree of insulin resistance is directly proportional to the accumulated free radicals. Selenium functions as an active site component of an antioxidant enzyme, glutathione peroxidase, and helps scavenge free radicals. In addition, an experimental study has shown that selenium provides activation by binding to insulin receptors and lowers blood sugar by increasing glucose uptake by cells.

According to all this information, we aimed to evaluate the effect of selenium on blood sugar regulation in pregnant patients.

DETAILED DESCRIPTION:
Pregnant patients with no known chronic disease / drug use and who had an oral glucose tolerance test between 24 and 28 weeks of gestation will be included in our study. The presence of one or more of the fasting blood glucose values ≥ 92, 1st Hour ≥ 180 and 2nd Hour ≥ 153 will be considered as gestational diabetes. Our patients diagnosed with gestational diabetes in the second step will be divided into two groups.

The first group will be started with diet only, the second group diet + 200 mcg selenium supplement per day. Patients will continue these treatments for 4 weeks, and at the end of 4 weeks, they will follow their fingertip blood sugar for 5 days (fasting, 1st hour satiety and 2nd hour satiety) while the treatment continues. In patients with gestational diabetes diagnosis, our targets for fingertip blood glucose follow-ups at home are fasting <95, 1st hour <140, 2nd hour <120.

The 5-day measurements of both groups will be averaged for fasting, 1st Hour and 2nd Hour, and it will be evaluated whether there is a significant difference in blood sugar regulation between the groups that take selenium supplements and those that do not.

ELIGIBILITY:
Inclusion Criteria:

* Presence of one or more of the values of fasting blood glucose ≥ 92, 1st hour ≥ 180 and 2nd hour ≥ 153 among pregnant patients for whom we had an oral glucose tolerance test between 24 and 28 weeks of gestation
* single pregnancy
* 18 to 45 years old

Exclusion Criteria:

* chronic disease (thyroid dysfunction, acute/chronic liver disease, acute/chronic kidney disease, hypertension )
* Patients with a diagnosis of insulin resistance or diabetes
* Those who use drugs other than iron, vitamin D and multivitamin support
* multiple pregnancy
* patients under 18 years old
* Patients over 45 years old

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
five day fasting glucose average | four weeks
  five-day fasting glucose average during treatment after one month of treatment
five-day first hour postprandial glucose average | four weeks
  five-day first hour postprandial glucose average during treatment after one month of treatment
five-day second hour postprandial glucose average | four weeks
  five-day second hour postprandial glucose average during treatment after one month of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided